CLINICAL TRIAL: NCT03515512
Title: A Phase I Study of IDH2 Inhibition Using Enasidenib as Maintenance Therapy for IDH2-mutant Myeloid Neoplasms Following Allogeneic Stem Cell Transplantation
Brief Title: IDH2 Inhibition Using Enasidenib as Maintenance Therapy for IDH2-mutant Myeloid Neoplasms Following Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Amir Fathi, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-022
Record Dates: First submitted 2018-04-23; First posted 2018-05-03 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia
Keywords: Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic | interventions — enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enasidenib (Experimental): Enasidenib will be administered orally once daily in 28-day cycles
  Interventions: Drug: Enasidenib

INTERVENTIONS:
Drug: Enasidenib — Enasidenib may help block the over production of IDH2, which when mutated, can overproduce metabolites and compounds that contribute to the growth of tumors and cancerous cells
  Other Names: idhifa

SUMMARY:
This research study is studying a targeted therapy drug as a possible treatment for IDH2 mutant acute myeloid leukemia or chronic myelomonocytic leukemia while undergoing hematopoietic stem cell transplantation.

The drug involved in this study is:

-Enasidenib.

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has approved enasidenib as a treatment option for some cancers, but not for the specific indication under study with this protocol.

Enasidenib is currently used to treat AML with an IDH2 mutation that has come back or has not improved after previous AML treatment. This study is examining whether or not enasidenib may be beneficial and well-tolerated as an agent to prevent the relapse of IDH2-mutated AML or other myeloid neoplasms after participants have undergone hematopoietic stem cell transplantation (HSCT). IDH2 is an enzyme that, when mutated, can overproduce metabolites and compounds that contribute to the growth of tumors and cancerous cells. Enasidenib may help block the over production of these substances.

There is an FDA-approved test available to detect IDH2 mutations in patients with AML, but for the purposes of participation in this clinical trial, an investigational test may be used to determine the presence of an IDH2 mutation.

In this research study, the investigators are:

* Looking for the maximum dose of enasidenib that individuals can take without experiencing severe side effects following HSCT.
* Looking at how often Graft-Versus-Host-Disease (GVHD) occurs in participants taking enasidenib. GVHD is a complication of transplant.
* Assessing the rates of relapse for participants taking enasidenib after HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of IDH2-mutant acute myeloid leukemia (AML), myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML).
* IDH2 mutations will include any IDH2 R140 or R172 alterations
* Eligibility and enrollment will be based on local IDH2 mutational testing performed at any center. The presence of an IDH2 mutation at the time of initial diagnosis or any other time thereafter is necessary and sufficient. The presence of an IDH2 mutation at time of enrollment is not necessary for the purposes of eligibility.
* Between the ages of 18 and 75 years
* Will undergo first allogeneic hematopoietic stem cell transplantation (HSCT) for their malignancy. Conditioning may have been either conventional myeloablative (MAC) or reduced intensity conditioning (RIC).
* HSCT Donor will be one of the following:

  * 5/6 or 6/6 (HLA-A, B, DR) matched related donor
  * 7/8 or 8/8 (HLA-A, B, DR, C) matched unrelated donor. Matching in the unrelated setting must be at the allele level.
  * Haploidentical related donor, defined as ≥ 3/6 (HLA-A, B, DR) matched --≥ 4/6 (HLA-A, B, DR) umbilical cord blood (UCB). Matching in the UCB setting is at the antigen level. Recipients may receive either one or two UCB units. In the case of 2 UCB units, both units must have been at least 4/6 matched with the recipient.
* ECOG performance status ≤ 2
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1000/µL without growth factor support (e.g. GCSF) in the previous 7 days
  * Platelet count ≥ 50,000/µL without transfusional support in the previous 7 days
  * AST (SGOT), ALT (SGPT) and Alkaline phosphatase < 3x institutional upper limit of normal (ULN)
  * Direct bilirubin < 2.0 mg/dL
  * Calculated creatinine clearance ≥ 40 mL/min (Cockcroft-Gault formula)
* LVEF must be equal to or greater than 50%, as measured by MUGA scan or echocardiogram
* Female patients of childbearing potential must have a negative pregnancy test, as measured by serum or urine testing
* The effects of enasidenib on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) during the entire study treatment period and through 6 months after the last dose of treatment
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior allogeneic hematopoietic stem cell transplants.
* Evidence of relapsed/recurrent/residual disease as assessed by bone marrow aspirate and biopsy performed within 42 days prior to study entry.
* History of other malignancy(ies) unless

  * the participant has been disease-free for at least 5 years and is deemed by the investigator to be at low risk of recurrence of that malignancy, or
  * the only prior malignancy was cervical cancer in situ and/or basal cell or squamous cell carcinoma of the skin
* Known diagnosis of active hepatitis B or hepatitis C
* Current or history of congestive heart failure New York Heart Association (NHYA) class 3 or 4, or any history of documented diastolic or systolic dysfunction (LVEF < 50%, as measured by MUGA scan or echocardiogram)
* Current or history of ventricular or life-threatening arrhythmias or diagnosis of long-QT syndrome
* Systemic infection requiring IV antibiotic or antifungal or antiviral therapy within 7 days preceding the first dose of study drug, or other severe infection
* Known dysphagia, short-gut syndrome, gastroparesis, or other condition(s) that limits the ingestion or gastrointestinal absorption of drugs administered orally
* Uncontrolled hypertension (systolic blood pressure [BP] > 180 mmHg or diastolic BP > 100 mmHg)
* QTc interval (i.e., Friderica's correction [QTcF]) ≥ 450 ms or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) at screening
* Concomitant receipt of the following sensitive CYP substrate medications that have a narrow therapeutic range (unless the participant can be transferred to other medications at least 5 half-lives prior to the start of study treatment): paclitaxel and docetaxel (CYP2C8), phenytoin (CYP2C9), S-mephenytoin (CYP2C19), thioridazine (CYP2D6), theophylline, and tizanidine (CYP1A2)
* Concomitant receipt of the breast cancer resistance protein (BCRP) transporter-sensitive substrate rosuvastain (unless the participant can be transferred to another medication at least 5 half-lives prior to the start of study treatment)
* Uncontrolled intercurrent illness that would limit compliance with study requirements.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with study drug. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 Days
  The maximum tolerated dose of Enasidenib in this patient population. The Maximum Tolerated Dose (MTD) is defined as the highest dose level at which 0 or 1 of six patients experiences a dose-limiting toxicity (DLT). MTD is determined using a standard 3 + 3 dose escalation cohort, where 3 participants will be enrolled on the starting dose of 50 mg daily and if no DLT is experienced after a full 28-day cycle, 3 additional participants will be enrolled at the next dose level of 100mg daily. If during any dose level, 1 patient out of 3 develops a DLT, then 3 additional patients will be added to that dose level. If 2 out of the 3 patients placed on any dose level experience a DLT, the preceding dose is considered MTD. If 1 out of 6 participants has a DLT, the next higher dose level will commence accrual. If ≥ 2 of 6 patients have a DLT, then the preceding dose will be considered MTD.
Number of participants with dose limiting toxicities (DLT) | 28 days
  Dose limiting toxicities are adverse events that occur during the first 28-day cycle that are considered serious enough to prevent an increase in the Enasidenib dose level. Adverse events are graded and documented per Common Terminology Criteria for Adverse Events (CTCAE 4).

SECONDARY OUTCOMES:
The number of participants with Enasidenib related adverse events | From the start of treatment until 30 days after the end of treatment, treatment may continue for up to 12 28-day cycles
  The number of participants with treatment related adverse events grouped by grade. Adverse events are assessed using Common Terminology Criteria for Adverse Events (CTCAE 4). Adverse events are considered to be related to treatment if they are deemed to be possibly, probably, or definitely related to treatment with Enasidenib by the investigator.
Cumulative incidence of acute GVHD | Cycle 1 days 1, 8, and 15; day 1 of every subsequent cycle (cycles are 28-days), up to 100 days after the start of treatment
  The cumulative incidence of acute graft versus host disease (GVHD). Acute GVHD is graded according to a composite grading of the clinical stages of skin rash, liver function, and intestinal tract function. Skin rash is assessed by the portion of the body covered by rash, liver function is assessed based on blood bilirubin levels, and intestinal track function is assessed based on the volume of diarrhea per day. The acute GVHD grade ranges from 1 to 4 with 1 representing less severe effects and 4 the most severe. The incidence represents the proportion of participants that experienced any grade acute GVHD.
Cumulative incidence of chronic GVHD | Cycle 1 days 1, 8, and 15; Day 1 of cycles 2-12 (1 cycle is 28-days), up to 1 year of total follow-up
  Cumulative incidence of chronic graft versus host disease (GVHD). cGHVD is assessed as per the National Institutes of Health consensus development project on criteria for clinical trials in cGVHD. cGVHD is graded as mild, moderate, or severe. The cGVHD grade is based on an aggregate score of different organ systems. The organ systems are graded from 0 to 3, with 0 being no-symptoms and 3 being the most severe symptoms. The cumulative incidence represents the proportion of participants that have any grade cGVHD.
  cGVHD Grade:
  * Mild: Involves only 1 or 2 organs or sites (except the lung), with no clinically significant functional impairment
  * Moderate: Involves at least 1 organ or site with clinically significant but no major disability or 3 or more organs or sites with no clinically significant functional impairment. A lung score of 1 will also be considered moderate cGVHD
  * Severe: Indicates major disability caused by cGVHD. A lung score of 2 will also be considered severe cGVHD
Plasma and marrow 2-hydroxyglutarate levels | Screening, cycle 1 days 8 and 15, day 1 of cycles 2 and 3, at the time of relapse, up to one year total follow-up
  Summary of the median 2-hydroxyglutarate levels at each time-point.
IDH clonal evolution via whole genome sequencing | Screening, cycle 1 days 8 and 15, day 1 of cycles 2 and 3, at the time of relapse, up to one year total follow-up
  Count summary of the specific Isocitrate dehydrogenase (IDH) mutations experienced by participants as assessed using whole genome sequencing.
IDH Mutational burden via next-generation sequencing | Screening, cycle 1 days 8 and 15, day 1 of cycles 2 and 3, at the time of relapse, up to one year total follow-up
  Summary of the number of mutations in the Isocitrate dehydrogenase (IDH) gene as assessed using next-generation sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Amir t Fathi, MD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Johns Hopkins Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fathi AT, Kim HT, Soiffer RJ, Levis MJ, Li S, Kim AS, Mims AS, DeFilipp Z, El-Jawahri A, McAfee SL, Brunner AM, Narayan R, Knight LW, Kelley D, Bottoms AS, Perry LH, Wahl JL, Brock J, Breton E, Ho VT, Chen YB. Enasidenib as maintenance following allogeneic hematopoietic cell transplantation for IDH2-mutated myeloid malignancies. Blood Adv. 2022 Nov 22;6(22):5857-5865. doi: 10.1182/bloodadvances.2022008632. PMID 36150050
- [Derived] Shallis RM, Podoltsev NA. Maintenance therapy for acute myeloid leukemia: sustaining the pursuit for sustained remission. Curr Opin Hematol. 2021 Mar 1;28(2):110-121. doi: 10.1097/MOH.0000000000000637. PMID 33394722